CLINICAL TRIAL: NCT01098019
Title: Efficacy and Safety of Xeomin for the Treatment of Notalgia Paresthetica
Brief Title: Treatment of Notalgia Paresthetica With Xeomin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-6014
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Notalgia Paresthetica
Keywords: Notalgia paresthetica; Xeomin; Botulinum Toxin A; Pruritus; Upper Back; Hyperpigmentation
MeSH Terms: conditions — Pruritus; Hyperpigmentation | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xeomin (Experimental): Each bottle of Xeomin will be reconstituted with 2 mL of NaCl 0.9 which will give a final concentration of 5 U of botulinum toxin A per 0.1 mL. The area affected will be injected with 0.1 mL at each 1-2 square cm for a maximum total dose of 200 units (4mL).
  Interventions: Drug: Xeomin
- Placebo (Placebo Comparator): Patients will receive 0.9% mL NaCl alone. The area affected will be injected with 0.1 mL at each 1-2 square cm for a maximum volume of 4 mL.
  Interventions: Drug: Placebo / Xeomin

INTERVENTIONS:
Drug: Xeomin — Patients will receive Xeomin only at Day 0.
  Other Names: Botulinum Toxin A
  Arms: Xeomin
Drug: Placebo / Xeomin — Patients will receive 0.9% mL NaCl alone at Day 0. After unblinding (at week 12) patients who were randomized to placebo will receive Xeomin.
  Other Names: Sodium Chloride; Saline
  Arms: Placebo

SUMMARY:
Patients will be randomized (1:1) to receive either injections of Xeomin in 0.9% NaCl or NaCl alone. Xeomin will be reconstituted with 2 mL of NaCl 0.9 which will give a final concentration of 5 U of botulinum toxin A per 0.1 mL. The area affected will be injected with 0.1 mL at each 1-2 cm2 for a maximum total dose of 200 units. Patients will be evaluated at Weeks 8, 12, 18 and 24. An unblinded pharmacist or designee will prepare placebo and Xeomin injections. Patients will be unblinded at the end of the week 12 visit. After unblinding (at week 12) patients who were randomized to placebo will receive Xeomin while patients initially randomized to Xeomin will not be injected. All patients will be seen for follow-up visits at Weeks 18 and 24. Efficacy in reducing pruritus will be measured with a 10 cm visual analogue score. This will be performed at Day 0, Week 8, Week 12, Week 18 and Week 24. Efficacy will also be measured by measuring the area of the hyperpigmented zone on the back. Safety will be evaluated with adverse events.

DETAILED DESCRIPTION:
Notalgia paresthetica is a common sensory neuropathy, affecting mainly the interscapular area especially the T2-T6 dermatomes. The characteristic symptom is pruritus on the upper back. It is occasionally accompanied by pain, paresthesia, hyperesthesia and a well circumscribed hyperpigmentation of the affected area. The correlation of notalgia paresthetica localization with corresponding degenerative changes in the spine suggest that spinal nerve impingement may be a contributing cause. Topical treatments such as corticosteroids, menthol, capsaicine and pramoxine are usually not very effective. Patients are very affected in their daily activities by this chronic condition and usually disappointed by the current available treatments.

A recent publication reports success in treating 2 patients with notalgia paresthetica with botulinum toxin A. In both cases a complete response for pruritus was noted. The major limitations of this publication are the small number of cases (two) and the fact that there was no control. The mechanism of action of botulinum toxin A in nostalgia paresthetica has not been investigated.

However the beneficial effects of botulinum toxin A on other diseases causing pruritus and pain has previously been reported. Botulinum toxin A has been shown to prevent the release of substance P, a well known mediator involved in pain and itch, and this may explain its efficacy in pruritic diseases. This proposal plans to study the efficacy and safety of botulinum toxin A (Xeomin) for the treatment of notalgia paresthetica in a randomized placebo controlled trial. Botulinum toxin A prevents the release of neuromediators such as acetylcholine. Botulinum toxin A has been used for many years to treat various disorders including blepharospasm, spasmodic torticollis, post stroke spasticity of the upper limbs, strabismus, palmar and axillary hyperhidrosis and wrinkles. This study will use Xeomin, a purified botulinum clostridium neurotoxin A that has recently been approved by Health Canada. Xeomin is currently approved for the treatment of blepharospasm, spasmodic torticollis and post stroke spasticity of the upper limbs.

A recent publication reported success in treating two patients with notalgia paresthetica with botulinum toxin A. In both cases a complete response of pruritus was noted. One patient was still symptom free after 18 months while the other patient had a mild resurgence of pruritus at 18 months. The major limitations of this publication are the small number of cases (two) and the fact that there was no control. The current proposal plans to study the efficacy and safety of botulinum toxin A for the treatment of notalgia paresthetica in a randomized placebo controlled trial. In this study Xeomin will be reconstituted and used according to the approved Canadian Product Monograph.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 75 years of age at the time of consent
* Presence of notalgia paresthetica, resistant to topical therapy, for at least one year and stable for the past 3 months prior to Day 0.
* Unless surgically sterile (or at least 1 year post-menopausal for women), or abstinent, patient (male or female) is willing to use an effective method of contraception for at least 30 days before Day 0 and until at least 12 months after the last drug administration. Effective method of contraception include:

  1. Condom with spermicidal foam or jelly, sponge with spermicidal foam or jelly, diaphragm with spermicidal foam or jelly
  2. Intra uterine device (IUD)
  3. Contraceptives (oral or parenteral)
  4. Nuvaring
  5. Vasectomy or vasectomised partner
  6. Surgically sterile or post-menopausal partner
  7. Same-sex partner
* Capable of giving informed consent; the consent must be obtained prior to any study related procedures.
* Negative urine pregnancy test (female of childbearing potential only)

Exclusion Criteria:

* Current Pregnancy of lactation
* Very mild notalgia paresthetica as defined by the absence of a clear zone of hyperpigmentation on the affected area on the back Severe notalgia paresthetica as defined by presence of excoriations, erosions or significant scarring in affected area on the back
* Use of any topical treatment on the affected area within 14 days of Day 0
* Use of botulinum toxin A within the past 12 weeks of Day 0
* Previous use of botulinum toxin A in the affected area on the back
* Use of systemic medication that can have an influence on pruritus such as antihistamines within 14 days of Day 0
* Use of systemic corticosteroids within 28 days of Day 0
* Hypersensitivity to Xeomin
* Generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert Eaton syndrome)
* Presence of infection on the affected area on the back

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Mean % difference in pruritus visual analog score (VAS). | 8 Weeks
  Changes from baseline in pruritus visual analogue score at Week 8 for patients randomized to Xeomin as compared to placebo

SECONDARY OUTCOMES:
Mean % difference in area of hyperpigmentation | 12 weeks
  Changes from baseline in area of hyperpigmentation on the affected zone of the back at Week 12 for patients randomized to Xeomin as compared to placebo
Mean % difference in area of hyperpigmentation | 24 weeks
  Changes from baseline in area of hyperpigmentation on the affected zone of the back at Week 24 as compared to baseline for patients randomized to Xeomin
Mean number of days before re-appearance of pruritus | 24 weeks
  Duration of efficacy as measured by changes from baseline in pruritus visual analogue score overtime for patients randomized to Xeomin
Mean global efficacy evaluated by investigator | 12 weeks
  Global efficacy of treatment as evaluated by the investigator at Week 12 for patients randomized to Xeomin as compared to placebo
Mean global efficacy evaluated by patient | 12 weeks
  Global efficacy of treatment as evaluated by patients at Week 12 for patients randomized to Xeomin as compared to placebo
Mean % difference in pruritus visual analogue score (VAS) | 12 weeks
  Changes from baseline in pruritus visual analogue score at Week 12 for patients randomized to Xeomin as compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Maari, MD, FRCPC, Principal Investigator — Innovaderm Research
Locations (1):
- Innovaderm Research Inc, Montreal, Quebec, Canada